CLINICAL TRIAL: NCT04754724
Title: Evaluation of GIMate Handheld Hydrogen Breath Monitor for Diagnosis of Lactose Malabsorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivante Health (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00107782
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-02

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIMate (Experimental): Individuals with suspected lactose intolerance who start with GIMate use first
  Interventions: Diagnostic Test: GIMate; Diagnostic Test: H2 Check
- H2 Check (Active Comparator): Individuals with suspected lactose intolerance who start with H2 Check use first
  Interventions: Diagnostic Test: GIMate; Diagnostic Test: H2 Check

INTERVENTIONS:
Diagnostic Test: GIMate — Use of GIMate to detect lactose malabsorption
Diagnostic Test: H2 Check — Use of H2 Check to detect lactose malabsorption

SUMMARY:
The goal of this study is to assess the performance of the Vivante Health GIMate Breathalyzer device in diagnosing lactose malabsorption.

DETAILED DESCRIPTION:
Lactose malabsorption is a common condition due to lactase deficiency which results in gastrointestinal symptoms for many which is termed lactose intolerance. Lactase is an enzyme occurring in the intestinal mucosa that hydrolyzes lactose into its constituent parts, galactose and glucose. The enzyme is normally present in neonates, however, for a majority of individuals in the world there is an inherited and irreversible reduction in enzyme activity as individuals age. Secondary lactose malabsorption can also occur when there is injury to the intestinal mucosa from a reversible condition such as infection.

The mechanism of hydrogen detection is based on undigested lactose in the colon being fermented by bacteria resulting in the production of hydrogen which is then partially absorbed into the bloodstream and ultimately exhaled by the lungs via the pulmonary circulation and gas exchange. Direct lactase activity can also be measured on tissue obtained through jejunal biopsy via endoscopy. This approach, however, is more invasive, costly, and potentially less reliable given issues relating to sampling bias

Current clinical hydrogen breath tests for diagnosis of lactose malabsorption are bulky and expensive for clinical providers to use and obtain. As a result, Vivante Health is testing how effective the GIMate device is in diagnosing lactose malabsorption as an alternative option.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female between 18 and 55 years of age (inclusive)
2. Able and willing to provide written consent and follow instructions to complete required study procedures (including dietary restriction) and questionnaires.
3. Self-reported or suspected history of lactose malabsorption or lactose intolerance

Exclusion Criteria:

Exclusion criteria:

1. History of prior gastrointestinal surgery
2. Self-reported history of any chronic gastrointestinal disease (examples include gastroesophageal reflux disease, celiac disease, Crohn's disease, ulcerative colitis, pancreatitis)
3. Self-reported history of endocrine or metabolic disease that may impact gastrointestinal or colonic function (examples include hyper/hypothyroidism, diabetes, etc)
4. Clinically significant cardiovascular, respiratory, renal, hepatic, hematologic, neurologic or psychiatric disease for which chronic therapy (prescription or non- prescription is required)
5. Self-reported history of allergic reaction to any drug or drug component
6. Antibiotic use within 28 days of lactose malabsorption test
7. Use of non-antibiotic prescription or OTC products (dietary or digestive supplements and laxatives) within 14 days of testing.
8. Self-reported use of nicotine-containing products or chronic secondhand smoke exposure within 14 days of testing.
9. Any other condition which in the Investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant.
10. Consumption of food after midnight on day of testing (within 12 hours) of testing or consumption of non-water beverage after midnight (or less than 8 hours) prior to testing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Positive percent agreement | immediately after the intervention
Negative percent agreement | immediately after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montalto M, Curigliano V, Santoro L, Vastola M, Cammarota G, Manna R, Gasbarrini A, Gasbarrini G. Management and treatment of lactose malabsorption. World J Gastroenterol. 2006 Jan 14;12(2):187-91. doi: 10.3748/wjg.v12.i2.187. PMID 16482616
- [Background] Gilat T, Russo S, Gelman-Malachi E, Aldor TA. Lactase in man: a nonadaptable enzyme. Gastroenterology. 1972 Jun;62(6):1125-7. No abstract available. PMID 5068338
- [Background] Wang Y, Harvey CB, Hollox EJ, Phillips AD, Poulter M, Clay P, Walker-Smith JA, Swallow DM. The genetically programmed down-regulation of lactase in children. Gastroenterology. 1998 Jun;114(6):1230-6. doi: 10.1016/s0016-5085(98)70429-9. PMID 9609760
- [Background] Labayen I, Forga L, Gonzalez A, Lenoir-Wijnkoop I, Nutr R, Martinez JA. Relationship between lactose digestion, gastrointestinal transit time and symptoms in lactose malabsorbers after dairy consumption. Aliment Pharmacol Ther. 2001 Apr;15(4):543-9. doi: 10.1046/j.1365-2036.2001.00952.x. PMID 11284784
- [Background] Shaw AD, Davies GJ. Lactose intolerance: problems in diagnosis and treatment. J Clin Gastroenterol. 1999 Apr;28(3):208-16. doi: 10.1097/00004836-199904000-00005. PMID 10192605
- [Background] Rezaie A, Buresi M, Lembo A, Lin H, McCallum R, Rao S, Schmulson M, Valdovinos M, Zakko S, Pimentel M. Hydrogen and Methane-Based Breath Testing in Gastrointestinal Disorders: The North American Consensus. Am J Gastroenterol. 2017 May;112(5):775-784. doi: 10.1038/ajg.2017.46. Epub 2017 Mar 21. PMID 28323273
- [Background] Peuhkuri K, Poussa T, Korpela R. Comparison of a portable breath hydrogen analyser (Micro H2) with a Quintron MicroLyzer in measuring lactose maldigestion, and the evaluation of a Micro H2 for diagnosing hypolactasia. Scand J Clin Lab Invest. 1998 May;58(3):217-24. doi: 10.1080/00365519850186607. PMID 9670345
- [Derived] Mathews SC, Templeton S, Taylor SK, Harris S, Stewart M, Raja SM. Evaluation of a Digital Handheld Hydrogen Breath Monitor to Diagnose Lactose Malabsorption: Interventional Crossover Study. JMIR Form Res. 2021 Oct 18;5(10):e33009. doi: 10.2196/33009. PMID 34544034